CLINICAL TRIAL: NCT02510937
Title: A Phase 1b, Multicenter, Open-label, Staggered-dose-escalation Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple Doses of CC-90001 for 3 Months in Patients With Pulmonary Fibrosis
Brief Title: Safety and PK Study of CC-90001 in Subjects With Pulmonary Fibrosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CC-90001-CP-003
Record Dates: First submitted 2015-07-27; First posted 2015-07-29 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Pulmonary Fibrosis
Keywords: pulmonary fibrosis; pharmacokinetic; pharmacodynamics; CC-90001; Safety
MeSH Terms: conditions — Pulmonary Fibrosis | interventions — CC-90001

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low dose CC-90001 (Experimental): Low dose (100 mg) CC-90001 administered orally once daily (QD) for 12 continuous weeks
  Interventions: Drug: CC-90001
- High dose CC-90001 (Experimental): High-dose (200 mg) CC-90001 administered orally Once Daily (QD) for 12 continuous weeks
  Interventions: Drug: CC-90001

INTERVENTIONS:
Drug: CC-90001

SUMMARY:
Participation in the study will last for 3months, with a 1 month screening phase.

DETAILED DESCRIPTION:
This is an open-label, staggered dose-escalation, cohort expansion study that will enroll subjects at multiple study sites in the United States of America (USA) and Australia. The study will consist of two treatment arms:

* Low dose (100 mg) CC-90001 administered orally once daily (QD) for 12 continuous weeks.
* High dose (200 mg) CC-90001 administered orally QD for 12 continuous weeks. The high dose (200 mg) CC-90001 arm will not start until at least three subjects complete a minimum of 2 weeks of low-dose CC 90001 and the low dose treatment arm is determined not to meet the study dose escalation stopping criteria (Figure 2).

Each subject will participate in a Screening (up to 4 weeks prior to treatment), a 12 week Treatment Phase, and a 4-week Follow-up visit. Subjects will be screened for eligibility. Subjects who meet all of the inclusion criteria and none of the exclusion criteria at Screening will return to the study site on Day 1 for assessments and to begin administration of a QD dose of CC 90001, according to the dose level in which the subject is enrolled. Three subjects will initially be enrolled to receive low dose CC-90001 (100 mg QD), and will be evaluated for all scheduled assessments through 12 weeks of treatment. Once a total of three subjects have completed the Week 2 visit, a decision to continue the study at the high dose level (200 mg QD) will be determined.

If the criteria for escalation to the high dose (CC-90001 200 mg QD) are met, the low dose (CC-90001 100 mg QD) subjects will remain on low dose (CC-90001 100 mg QD) and six additional subjects will be enrolled at the high dose level (CC-90001 200 mg QD). If one of the three subjects at the low dose (CC-90001 100 mg QD) experiences an event that meets the individual subject dose stopping criteria, another three subjects will be enrolled in the low dose arm. Dose escalation to the high dose (CC-90001 200 mg QD) will not occur if two or more of the six subjects meet the individual subject dose stopping criteria. All subjects (low and high dose) will remain on CC-90001 for a total of 12 weeks unless an individual subject experiences an event that meets any of the individual subject stopping criteria. In addition, the dose of CC-90001 may be reduced CC-90001 200 mg QD to CC-90001 100 mg QD) for an individual who meets any of the individual subject dose reduction criteria. If two or more subjects in the high dose (CC-90001 200 mg QD) arm experience an event that meets the individual stopping criteria, the 100 mg QD dose arm may be repeated in three additional subjects, or the study may be stopped.

Study visits will occur at Screening, Day 1, and Weeks 1, 2, 3, 4, 6, 8, 10, 12, and 16 (a Follow-up visit). Blood and urine samples will be collected at specified times for clinical safety laboratory assessments, pharmacokinetic analysis (how the drug affects the body), and pharmacodynamic analysis (how the body affects the drug). Safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Potential subjects must satisfy all of the following criteria to be enrolled into the study:

  1. Subject ≥ 18 years of age.
  2. Documented clinical diagnosis of a fibrotic lung disease supported by at least one of the following:

     1. Usual interstitial pneumonia (UIP) pattern based on high-resolution computed tomography (HRCT).

        OR
     2. Nonspecific interstitial pneumonia (NSIP) pattern based on HRCT. OR
     3. A documented fibrotic NSIP on surgical lung biopsy. OR
     4. A documented UIP pattern on surgical lung biopsy. The underlying etiology of the fibrotic lung disease may be of any cause, including, but NOT LIMITED TO any of the following: Connective tissue disease associated interstitial lung disease, idiopathic pulmonary fibrosis (IPF), environmental or chemical-related pulmonary fibrosis, other forms of interstitial pulmonary fibrosis, Hermansky-Pudlak syndrome.
  3. Must understand and voluntarily sign a written Informed Consent Form prior to any study-related procedures being performed.
  4. Must be able to communicate with the Investigator, understand and comply with the requirements of the study, and agree to adhere to restrictions and examination schedules.
  5. Asparate Aminotransferase (AST) or serum glutamic-oxaloacetic transaminase within limits of normal.
  6. Alanine Aminotransferase (ALT) or serum glutamic pyruvic transaminase within limits of normal.
  7. Total bilirubin and International Normalized Ratio (INR) within limits of normal.
  8. No clinically significant laboratory test results as determined by the Investigator.
  9. Male subjects agree to use barrier contraception NOT made of natural (animal) membrane (eg, latex or polyurethane condoms are acceptable) when engaging in sexual activity with a female of childbearing potential (FCBP) while on CC 90001 and for at least 28 days after the last dose of study medication. A FCBP is defined as a sexually mature female who has not undergone a hysterectomy or bilateral oophorectomy or who has not been naturally postmenopausal for at least 24 consecutive months (ie, who has had menses at any time in the preceding 24 consecutive months).
  10. All FCBPs must have a negative pregnancy test at Screening and Day 1. Any FCBP who engages in activity in which conception is possible must use two forms of contraception simultaneously while on CC-90001 and for at least 28 days after taking the last dose of CC-90001: one highly effective form (ie, hormonal, intrauterine device, tubal ligation, vasectomized partner) and one additional form (latex condom or any nonlatex condom NOT made of natural [animal] membrane [eg, polyurethane], diaphragm, sponge). If one highly effective form of contraception cannot be used, then two forms of barrier contraception must be used, ie, latex condom or any nonlatex condom NOT made out of natural (animal) membrane [eg, polyurethane] with either of the following: sponge with spermicide or diaphragm with spermicide.
  11. Female subjects that are postmenopausal (defined as 24 months without menses before Screening, with an estradiol level of < 30 pg/mL and FSH level of > 40 IU/L at Screening).

Exclusion Criteria:

* Potential subjects will be excluded from enrollment if any of the following occur:

  1. Exposed to an investigational drug (new chemical entity) within 30 days preceding the first dose of CC-90001 administration, or five half-lives of that investigational drug, if known (whichever is longer).
  2. Subjects who are part of the clinical staff personnel or family members of the study site staff.
  3. Screening forced vital capacity (FVC) < 40% predicted.
  4. Screening lung diffusion capacity (DLco) < 20% predicted.
  5. Any condition other than pulmonary fibrosis that is likely to result in the subject's death or increases the risk of death within a year from signing the ICF.
  6. Known clinical diagnosis of pulmonary arterial hypertension that currently requires treatment.
  7. Subjects with cystic fibrosis, active aspergillosis, active tuberculosis, or other serious concomitant respiratory disorder other than pulmonary fibrosis, as determined by the Investigator. Subjects with reactive airway disease, chronic obstructive pulmonary disease, and asthma may be included as long as, in the opinion of the Investigator, fibrosis is the major contributing factor to the subject's respiratory disorder.
  8. Use of any cytotoxic agents within 4 weeks of dosing.
  9. Currently being administered any targeted therapy for pulmonary fibrosis and not on a stable dose for ≥ 6 weeks duration prior to first study dosing (potential subjects should be excluded if a dose increase is planned during the study period).
  10. Use of Esbriet® (pirfenidone) or Ofev® (nintedanib) within 30 day prior to first dose.
  11. Currently being administered statins (HMG-CoA reductase inhibitors) and not on a stable dose for ≥ 6 weeks duration prior to first study dosing (potential subjects should be excluded if a dose increase is planned during the study period).
  12. Taking medications that are substrates of the transporters P-gp, BCRP, OAT3, OATP1B1, OATP1B3, and OCT2 and have a narrow therapeutics index (eg, P-gp substrate digoxin).
  13. Use of acetaminophen (paracetamol) at a dosage > 3 grams per day within 2 weeks of first study dosing.
  14. Use of niacin at a dosage > 2 grams/day within 2 weeks prior to first study dosing.
  15. Any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study.
  16. History of recurrent bacterial infections (at least three major infections resulting in hospitalization and/or requiring intravenous antibiotic treatment within the past 2 years)
  17. History of Human Immunodeficiency (HIV), Hepatitis B Virus (HBV), or Hepatitis C Virus (HCV). Subjects treated for HCV who have a sustained virologic response of 6 months following final HCV treatment can be included.
  18. History of active malignancy within 5 years prior to signing the ICF, excluding nonmelanoma skin cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-08-05 (Actual); Primary Completion 2017-02-06 (Actual); Study Completion 2017-02-06 (Actual)

PRIMARY OUTCOMES:
Adverse Events (AEs) | up to 16 weeks
  Number of subjects with adverse events
Dose interruptions, reductions, and discontinuation | up to 16 weeks
  Number of subjects experiencing dose interruptions, reductions, and discontinuation of CC-90001 secondary to an AE
Complete PEs | up to 16 weeks
  Complete Physical Examinations
Clinical laboratory assessments | up to 16 weeks
  Clinical laboratory assessments
Vital sign measurements | up to 16 weeks
  Heart rate (HR), respiratory rate, blood pressure (BP), and body temperature
12-lead ECGs | up to 16 weeks
  12-lead ECGs
Urine pregnancy tests | up to 16 weeks
  Urine pregnancy tests
Concomitant medications and procedures | up to 16 weeks
  Concomitant medications and procedures

SECONDARY OUTCOMES:
CC-90001 plasma concentrations | up to 16 weeks
  CC-90001 plasma concentrations collected sparsely and measured using a validated liquid chromatography tandem mass spectrometry assay
Population-based PK | up to 16 weeks
  Population-based PK approach as appropriate for the following parameters (at a minimum, but not limited to): apparent clearance; apparent central volume of distribution; first-order rate of absorption; disease as a covariate may be explored in the population PK analysis-the derived PK parameters such as Cmax and AUC may be also determined based on the population PK model as appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Ed O'Mara, MD, Study Director — Celgene Corporation
Locations (6):
- United States (4):
  - Tampa General Hospital, Tampa, Florida
  - LaPorte County Institute for Clinical Research, Inc, Michigan City, Indiana
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
- Australia (2):
  - The Prince Charles Hospital, Chermside
  - St. Vincent's Hospital- Sydney, Darlinghurst